CLINICAL TRIAL: NCT01765634
Title: Mesenchymal Stem Cells From Third-party Donors for Treatment of Refractory Acute Graft-versus-host Disease
Brief Title: Mesenchymal Stem Cells for Treatment of Refractory Acute Graft-versus-host Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Sun Yat-sen University (Other); Peking University People's Hospital (Other); Guangdong Provincial People's Hospital (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); Southern Medical University, China (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Guangzhou First People's Hospital (Other); Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFH-MSCs-aGVHD-2013
Record Dates: First submitted 2013-01-05; First posted 2013-01-10 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Acute Graft-versus-host Disease
Keywords: Hematopoietic Stem Cell Transplantation; Mesenchymal Stem Cells; Acute Graft-versus-host disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesenchymal stem cells (Experimental): Mesenchymal stem cell group refers to treatment with mesenchymal stem cells (1×10^6 cells/kg, intravenously)each week, four times for a cycle
  Interventions: Biological: Mesenchymal stem cells
- Non-mesenchymal stem cells (Experimental): Non-mesenchymal stem cell group refers to treatment with other second line drugs
  Interventions: Biological: Non-mesenchymal stem cells

INTERVENTIONS:
Biological: Mesenchymal stem cells — Mesenchymal stem cells will be intravenously infused via a central venous catheter(at a dose of 1×10^6 cells/kg, over 15 min) each week, four times for a cycle.
  Other Names: Mscs
  Arms: Mesenchymal stem cells
Biological: Non-mesenchymal stem cells — Other second line drugs are taken.
  Other Names: Non-MSCs
  Arms: Non-mesenchymal stem cells

SUMMARY:
The purpose of this study is to evaluate the utility of treating patients experiencing refractory acute graft-versus-host disease with ex-vivo-expanded BM-drived mesenchymal stem cells from third-party donors. The objective was to evaluate the effect and safety of such treatment on refractory acute graft-versus-host disease.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation(allo-HSCT) can cure many hematologic diseases. Although great progress has been made in the prevention and treatment of side effects associated with transplantation,acute graft-versus-host disease(aGVHD) remains an important complication that occurs in 35-80% patients. The mortality of aGVHD is positively correlated with its severity. At present, glucocorticoids is still the first line treatment of aGVHD. If glucocorticoids treatment is ineffective, second line drugs would be taken, such as tacrolimus(FK506), mycophenolate mofetil (MMF)and antithymocyte globulin (ATG). However, no method could be continuously effective. The effective rates of second line treatment to aGVHD is only about 60%. The effective rates and prognosis of refractory aGVHD are even worse.

Mesenchymal stem cells (MSCs) are a form of multipotent adult stem cells that can be isolated from bone marrow (BM), adipose tissue, and cord blood. Clinical applications of human MSCs are evolving rapidly with goals of improving hematopoietic engraftment, preventing and treating GVHD after allo-HSCT and so on. However, the efficacy of treatment of refractory aGVHD using expanded BM-derived MSCs from a third-party donor is rarely reported. If such treatment could be shown to be effective and safe, BM-derived MSCs could potentially be used as an universal donor material. This would have a major impact because the generation of donor-specific MSCs is time-consuming, costly, and often impractical if the clinical status of a patient is urgent.

In the present study, the investigators will prospectively evaluate the efficacy and safety of ex-vivo-expanded BM-derived MSCs from third-party donors in treating patients with refractory aGVHD.

ELIGIBILITY:
Inclusion Criteria:

* A patient age of 12-65 years
* Recipients of allogeneic hematopoietic stem cell transplantation
* Patients with refractory aGVHD
* On a voluntary basis, patients are divided into MSCs and Non-MSCs group
* Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The efficacy of treatment for refractory aGVHD | 1 year
  The response criteria include complete response (CR), part response (PR), stable disease(SD) and progressive disease(PD). CR:aGVHD symptoms and signs disappear; PR:aGVHD symptoms and signs improve; SD:aGVHD symptoms and signs remain (without improvement or deterioration);PD: aGVHD symptoms and signs deteriorate.

SECONDARY OUTCOMES:
acute and late toxic side effects of MSCs treatment | 1 year
  Toxic side effects of treatment includes acute toxicity and late side effects. Acute toxicity principally involves the heart,live and kidney. Late toxic side effects involves principally the development of secondary tumors and relapse of the primary disease.

OTHER OUTCOMES:
infections | 1 year
  Infections will be mainly focused within the first 100 days after MSCs treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Le Blanc K, Frassoni F, Ball L, Locatelli F, Roelofs H, Lewis I, Lanino E, Sundberg B, Bernardo ME, Remberger M, Dini G, Egeler RM, Bacigalupo A, Fibbe W, Ringden O; Developmental Committee of the European Group for Blood and Marrow Transplantation. Mesenchymal stem cells for treatment of steroid-resistant, severe, acute graft-versus-host disease: a phase II study. Lancet. 2008 May 10;371(9624):1579-86. doi: 10.1016/S0140-6736(08)60690-X. PMID 18468541
- [Background] von Bonin M, Stolzel F, Goedecke A, Richter K, Wuschek N, Holig K, Platzbecker U, Illmer T, Schaich M, Schetelig J, Kiani A, Ordemann R, Ehninger G, Schmitz M, Bornhauser M. Treatment of refractory acute GVHD with third-party MSC expanded in platelet lysate-containing medium. Bone Marrow Transplant. 2009 Feb;43(3):245-51. doi: 10.1038/bmt.2008.316. Epub 2008 Sep 29. PMID 18820709